CLINICAL TRIAL: NCT07350694
Title: Engagement of coMmunity Through Participatory Learning and Action for cOntrol and preVEntion of Type II Diabetes and Its Risk Factors [EMPOWER-D-Afg]: Feasibility Trial in Rural Kabul-Afghanistan
Brief Title: Engagement of coMmunity Through Participatory Learning and Action for cOntrol and preVEntion of Type II Diabetes and Its Risk Factors
Acronym: EMPOWER-D-Afg
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HealthNet Transcultural Psychosocial Organization (Other)
Collaborators: University of York (Other); Khyber Medical University Peshawar (Other); National Institute for Health Research, United Kingdom (Other Government); Aga Khan University (Other)
Responsible Party: Principal Investigator, Sayed Murtaza Sayed Murtaza Sadat Hofiani, Research coordinator, HealthNet TPO, HealthNet Transcultural Psychosocial Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HealthNet TPO, A-12-24-464; NIHR 203248 (Other Grant/Funding Number: National Institute of Health and Care Research)
Record Dates: First submitted 2025-11-16; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Type 2; Type II Diabetes Mellitus
Keywords: Community-Based Participatory Research; Participatory Learning and Action Research; Type II Diabetes Mellitus; Intermediate hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Two-arm parallel study design would be used (Intervention and Control Arms)
  Study Site Details:
  1. province: Kabul
  2. districts: (District 1 and 2)
  4 clusters: (villages) 2 cluster (intervention arm) and 2 clusters (control arm)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLA Intervention group (Experimental): Participatory Learning and Action (PLA) sessions adapted from the D-MAGIC trial (Bangladesh). The PLA intervention will be delivered to community members with type II diabetes to improve diabetes-related outcomes. Sessions will be group-based, lasting approximately 2-3 hours each. Participants in this arm will be followed and evaluated 10 months after the start of the intervention using a structured, validated, literature-based endline assessment checklist to assess feasibility and outcomes.
  Interventions: Behavioral: PLA
- Usual care (control) group (No Intervention): Participants in the control arm will receive standard practice (usual care) and comprehensive information about the project but will not receive the PLA intervention.

INTERVENTIONS:
Behavioral: PLA — An PLA based intervention would be carried out to prepare the individuals with TIIDM. The intervention would be carried out for a tentative time of 2 to 3 hours to educate the community. The study participants would be evaluated after completion of 10 months of the intervention. A structured, validated and literature-based end line assessment checklist will be devised to assess the feasibility of the intervention.
  Other Names: Participatory Learning and Action
  Arms: PLA Intervention group

SUMMARY:
This project aims to adapt, implement, and evaluate PLA based intervention in Rural Kabul, Afghanistan for TIIDM prevention and control.

DETAILED DESCRIPTION:
This approach centres on adapting, implementing, and evaluating a Participatory Learning and Action (PLA) based intervention for the prevention and control of Type II Diabetes. Mellitus (TIIDM). TIIDM is one of the fastest-growing health emergencies globally, affecting an estimated 589 million adults, with projections for 2050 indicating a 45% increase in diabetes. Approximately 80% of people with TIIDM live in low- and middle-income countries (LMICs), placing further strain on already overburdened health systems.

Afghanistan shows similarly concerning trends, with an age-standardised diabetes prevalence of 11.7%, affecting 1.93 million adults in 2024 and projected to rise to 4.76 million by 2050, with 71.4% remaining undiagnosed. Prevalence rises sharply with age and varies by province for example, approximately 11% in Kabul, 11.8% in Nangarhar, and over 22% in Kandahar. These figures highlight the urgency of developing culturally appropriate and evidence-based interventions to prevent and control diabetes in Afghan communities.

The intervention draws on evidence from the "Community groups or mobile phone messaging to prevent and control type 2 diabetes and intermediate hyperglycaemia in Bangladesh (DMagic)" trial, which proved effective in rural Bangladesh. However, PLA-based interventions have yet to be tested in rural Afghan communities. Recognizing the distinct sociocultural context, geopolitical and health system challenges in rural Kabul, Afghanistan, a feasibility trial will be carried out in selected rural sites of Kabul Province.

This feasibility trial will evaluate the adaptability and implementation of the intervention within Afghanistan's context. By applying evidence-based practices and fostering meaningful community participation through PLA, the initiative aims to improve social and behavioural determinants of health, enhance diabetes prevention and control, and create a model for addressing other non-communicable diseases in Afghan communities.

ELIGIBILITY:
Inclusion Criteria:

* For intervention phase: Individuals aged 20 years and above. For baseline and endline assessments (before and after the intervention): Individuals aged 30 years and above.
* Participants residing in the randomized clusters of Kabul, Afghanistan Individuals willing to participate in the study and provide consent.
* All individuals with normoglycemia, intermediate hyperglycaemia, and diabetes are encouraged to participate.
* Participants who can attend the scheduled meetings and interventions as per the study protocol.

Exclusion Criteria:

* For Intervention phase: Individuals below the age of 20 years. For baseline and endline assessments (before and after the intervention): individuals below the age of 30 years.
* Individuals unwilling to provide consent for participation.
* Participants with reported health conditions that may hinder their active involvement in the study.
* Individuals with non-compliance with research protocols

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both Genders (Male and Female)
Enrollment: 250 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
To culturally adapt PLA-based intervention (D-Magic) for primary prevention and control of TIIDM in rural communities of Afghanistan | 10 months
  The outcome will measure the total number of Participatory Learning and Action (PLA) meetings conducted according to the adapted PLA manual. A total of 40 sessions are planned across four PLA groups (two male groups and two female groups), with 10 sessions per group. This measure will report the number of sessions completed as scheduled.
To test the feasibility of the culturally adapted PLA-based intervention (D-Magic) | 12 months
  Definition: Feasibility is measured by the number of participants attending PLA meetings, reflecting successful delivery and engagement.
  Measurement: Number of attendees (N) and proportion (%) of invited participants attending at least one PLA session.
To test the acceptability of the culturally adapted PLA-based intervention (D-Magic) | 12 months
  Definition: Acceptability is assessed by participant retention across PLA meetings, reflecting continued engagement and satisfaction with the intervention.
  Measurement: Number of participants completing the series of PLA meetings (N) and proportion (%) retained.

SECONDARY OUTCOMES:
To estimate the inter-correlation coefficient to inform future adjustment of sample size | 6 months
  The intra-cluster correlation coefficient (ICC) will be estimated to assess within-cluster similarity. Both measures will provide essential parameters for designing a future full-scale rural trial.
To identify and examine potential Barriers to Implementation of the PLA-Based Intervention | 12 months
  Definition: Barriers to implementing the PLA-based intervention, including logistical, operational, cultural, and community-related challenges.
  Measurement: Identified and assessed through process evaluation using supervisory checklists, supervision reports, meeting minutes, participant feedback, and qualitative data from FGDs and IDIs. Each barrier will be coded and categorized into predefined domains.
  Unit of Measure: Number of unique barriers identified in each category (count) and descriptive summaries.
To identify and examine potential facilitators of Implementation of the PLA-Based Intervention | 12 months
  Definition: Factors that facilitate successful implementation of the PLA-based intervention, including community engagement strategies, mobilizer practices, and contextual supports.
  Measurement: Identified and assessed through process evaluation using the same tools: supervisory checklists, supervision reports, meeting minutes, participant feedback, and qualitative data from FGDs and IDIs. Facilitators will be coded and categorized into predefined domains.
  Unit of Measure: Number of unique facilitators identified in each category (count) and descriptive summaries.
To assess the frequency of Type 2 Diabetes and Intermediate Hyperglycaemia | 12 months
  Type 2 diabetes and intermediate hyperglycaemia will be assessed at baseline and endline of the intervention using biochemical measurements, including fasting blood glucose and HbA1c, based on standard clinical cut-off values.
  Additional cardiometabolic risk factors will be assessed at baseline and endline, including anthropometric measurements (weight and height) and selected behavioural factors collected using standardised questionnaires (Food Frequency Questionnaire, Physical Activity Questionnaire and WHOQOL-BREF). Sociodemographic information will be collected using a structured case report form. Outcomes will be reported as counts and percentages only.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Rahman Shahab, MPH, Principal Investigator — Deputy Country Director, HealthNet TPO, Afghanistan
Locations (1):
- HealthNet TPO, Afghanistan, Kabul, Kabul, Afghanistan

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in the stated study area after its proper monitoring. Data or samples shared will be coded, with no Protected Health Information included. Prior permission of the investigators, participants and concerned departments will be obtained.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 12 months after article publication
Access Criteria: Access can be requested by qualified researchers through proper approval of the investigators.

REFERENCES:
- See also: Afghanistan, Diabetes country report 2011 - 2050, Diabetes Atlas, International Diabetes Federation, 2025. Data extracted from — https://diabetesatlas.org/data-by-location/country/afghanistan/